CLINICAL TRIAL: NCT03518385
Title: Does the Presence of Intracavitary Fluid During Hormonal Stimulation for IVF Depends on the Position of C-section-scar?
Brief Title: Intracavitary Fluid and Position of C-section-scar
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 1802-ABU-018-HF
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Fluid Uterus
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with intracavitary fluid: to evaluate the correlation between the presence of intracavitary fluid during hormonal stimulation for IVF depending on the position of C-section-scar and the presence of an isthmocele, this group patients will have intracavitary fluid.
  Interventions: Diagnostic Test: ultrasound,transvaginal scan
- Patients without intracavitary fluid: to evaluate the correlation between the presence of intracavitary fluid during hormonal stimulation for IVF depending on the position of C-section-scar and the presence of an isthmocele, in this group patients will not have intracavitary fluid.
  Interventions: Diagnostic Test: ultrasound,transvaginal scan

INTERVENTIONS:
Diagnostic Test: ultrasound,transvaginal scan — The presence of fluid in the uterine cavity during hormonal stimulation.

SUMMARY:
Does the presence of intracavitary fluid during hormonal stimulation for IVF depends on the position of C-section-scar ?

DETAILED DESCRIPTION:
To evaluate the correlation between the presence of intracavitary fluid and the position of the C-section-scar in relation to the uterine fundus and the inner cervical os.

To this end, we will compare measured variables, in patients with intracavitary fluid and without intracavitary fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patients above an age of 18 years.
* Patients performing IVF treatment.
* One or multiple C-sections.
* C-scar region visible during trans-vaginal scan.

Exclusion Criteria:

* Patients who were IUD carriers in the last 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients undergoing IVF treatment in the IVI Middle East Clinic Abu Dhabi and Dubai, due to secondary infertility and delivery with at least one previous C-section.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Presence/Absence of ICF | 1 year and 6 months
  to evaluate the correlation between the presence of intracavitary fluid and the position of the C-section-scar in relation to the inner cervical os, during hormonal stimulation for IVF.

SECONDARY OUTCOMES:
Thickness of fluid accumulation in the cavity | 1 year and 6 months
  Presence or Absence of ICF

CONTACTS AND LOCATIONS:
Overall Officials: Human Fatemi, MD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bij de Vaate AJ, Brolmann HA, van der Voet LF, van der Slikke JW, Veersema S, Huirne JA. Ultrasound evaluation of the Cesarean scar: relation between a niche and postmenstrual spotting. Ultrasound Obstet Gynecol. 2011 Jan;37(1):93-9. doi: 10.1002/uog.8864. PMID 21031351
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Background] Chien LW, Au HK, Xiao J, Tzeng CR. Fluid accumulation within the uterine cavity reduces pregnancy rates in women undergoing IVF. Hum Reprod. 2002 Feb;17(2):351-6. doi: 10.1093/humrep/17.2.351. PMID 11821277
- [Derived] Lawrenz B, Melado L, Garrido N, Coughlan C, Markova D, Fatemi H. Isthmocele and ovarian stimulation for IVF: considerations for a reproductive medicine specialist. Hum Reprod. 2020 Jan 1;35(1):89-99. doi: 10.1093/humrep/dez241. PMID 31885047
- See also: Rise in number of C-section deliveries. — http://gulfnews.com/news/uae/health/rise-in-number-of-c-section-deliveries-1.1787773